CLINICAL TRIAL: NCT00745537
Title: Teens--Building Options and Opportunities for Moms
Brief Title: T- BOOM Teens--Building Options and Opportunities for Moms
Acronym: T-BOOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Katherine Wisner, Professor of Psychiatry, University of Pittsburgh
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: B7473
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Postpartum Major Depression
Keywords: postpartum major depression; adolescent mothers; telephone depression care management; barriers to depression care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adolescent Mother (Experimental): aged less than 17 years old and recently gave birth
  Interventions: Other: repeated mood measures and phone depression care management

INTERVENTIONS:
Other: repeated mood measures and phone depression care management — The adolescent mothers will be assigned a depression care management who will support the mother in making choices about depression treatment, educate about treatment options, discuss barriers and solutions, counsel to comply with treatment recommendations, and assisted to problem-solve if failure to respond occurs.

SUMMARY:
Postpartum depression (PPD) is depression that occurs shortly after the mother delivers her baby. Mothers with postpartum depression may feel sad mood, low motivation or stress; some may have problems caring for their new baby. Successful depression treatment involves early screening and detection of postpartum depression and early access to treatment services.

The purpose of this study is to evaluate the effectiveness of a telephone-based depression screening and care management program for postpartum women. We will evaluate the: 1) how often (frequency) young mothers develop symptoms of depression 4 to 6 weeks after birth, 2) how quickly (timeliness) young mother receive treatment and how effective (adequacy) are the treatments for the symptoms of postpartum depression, 3) the effects of depression care support on young mothers' symptoms and their ability to function at 3, 6 and 12 months after entering the study, 4) visits to the pediatrician or nurse practitioner (preventive health services) during their baby's first year of life, and 5) cost and cost savings associated with depression care management.

DETAILED DESCRIPTION:
Depression during the perinatal period is a major public health concern. Postpartum depression (PPD) causes personal and family suffering at a time when adaptation to parenthood is critical. Successful interventions for treating depression in medical settings have been framed by a chronic disease management model. The key ingredient to success is a dedicated care manager who provides education and support to patients, actively coordinates care, and thereby improves treatment outcomes for patients. Compared to interventions in medical office settings, telephone care management positioned at the level of the health plan offers a systematic and efficient mechanism for ongoing treatment support of women with PPD, particularly in a geographically dispersed population.

We propose to conduct a comprehensive project to improve treatment outcomes for depressed postpartum women through adaptation of the depression care management model used in primary care settings. The major components are: 1) depression screening in a population of postpartum adolescents, 2) depression education for all who screen positive, 3) a diagnostic interview to evaluate for depressive disorders in mothers who score above and below a defined threshold on the screening instrument, 4) telephone-based care management intervention, and 5) longitudinal evaluation across the first year post-birth for depression and maternal and child public health outcomes. Focus groups will precede the major study components. A focus group of adolescent mothers will inform the investigators about the barriers to depression care management that encompass resource needs, acceptability of interventions to cope with stress or depression, and access to care. A separate focus group of community professionals of representatives from agencies or groups that provide community supports and health services will be used to explore the perceptions of barriers to care for new adolescent mothers. All participants in this project will be eligible for mental health services through their health plans that serve Medicaid and commercial members.

We plan to identify 125 child or adolescent new mothers with PPD. The child or adolescent new mothers will be assigned to depression care management. They will be supported in making choices about depression treatment (after receiving education about options), encouraged to access their preferred treatment (through the direct discussion of barriers and solutions), counseled to comply with treatment recommendations, and assisted to problem-solve if failure to respond occurs. All participants will have systematic evaluations at 3, 6, and 12 months post-birth. Outcomes include not only maternal depressive symptom levels but also functional and public health outcomes for mothers, families, and infants. We have developed a multi-disciplinary team with expertise in clinical research with depressed and minority women and health services to address these needs.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent mothers age < 17 years 364 days at birth of index infant
* Live born infants
* Parents/guardian of the young mother must be available and competent to provide consent to the enrollment of the young mother
* The young mother may provide assent for her own enrollment.
* Ethical need for awareness of the possible risks, benefits and alternatives to enrollment in this study.
* Mothers with an EPDS>/=10 or CES-D>/=16 (suggest increased risk for major depression)
* Mothers with major depressive disorder (MDD) regardless of their EPDS or CES-D scores. These are patients with high risk for severe recurrence of depressive symptoms in the postpartum. We will assess their outcomes in this study.
* Adolescent mothers with an EPDS<10 OR CES-D<16 (screen negative) without MDD will be interviewed by phone with the KIDDIE-SADS mood screen to screen for all categories of major diagnoses AND the Mood Disorders Module

Exclusion Criteria:

* No access to a telephone Screening and depression care management are accomplished by phone; mothers with no phone are referred to Magee social work for other services
* NON-English-speaking Measures are in English
* The multiple questionnaires and measures are in English

Ages: 10 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2008-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Severity of PPD will be assessed with the Children's Depression Rating Scale (CDRS). | Trained interviewers will complete the CDRS at baseline, 3, 6, and 12 months postpartum.
Edinburgh Postnatal Depression Scale | Baseline, 3, 6, and 12 months
Center for Epidemiologic Studies of Depression instrument (CES-D) | Baseline, 3, 6 and 12 months

SECONDARY OUTCOMES:
A specific measure of functioning at school or work and with peers, the Children's Global Assessment of Functioning (C-GAS) will be obtained. | baseline, 3, 6, and 12 months
The Social Function-12 (SF-12; Ware et al., 1993) is the most widely used measure of health-related functioning. | baseline, 3, 6, 12 months
The Inventory of Functional Status after Birth (IFSAC) was used in studies of postpartum women to measure the woman's readiness to assume infant care and resume usual activities (Fawcett et al., 1988). | baseline, 3, 6 and 12 months
To assess the mother-infant relational quality, the Gratification in the Maternal Role (GRAT) is a 14-item checklist in which women rate each item on a 5 point scale (Mercer, 1985). | Baseline, 3, 6 and 12months

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L Wisner, M.D., Principal Investigator — 3811 O'Hara Street, Oxford 410, Pittsburgh, PA 15123
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States